CLINICAL TRIAL: NCT05267353
Title: School of Nursing, College of Medicine, National Taiwan University
Brief Title: Develop and Test the 'Multi-Faced Continuous Exercise Program' in Operable Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 201209068RIC
Record Dates: First submitted 2022-02-11; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; neck dissection; exercise intervention; quality of life; physical function
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: A pre- and post- study design was used to recruit patients. Data collection for usual care (control) group was completed before recruitment of exercise (intervention) group.
Masking Description: Blindness is difficult to perform, all patients are treated at the same hospital, and contamination of the control group is easy. Hence, a pre- and post- study would be conducted and patients in exercise group were recruited based on gender and type of neck dissection in control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): All patients received care as usual. Patients receive wound care and pain management post-surgery. Before RT, generally advising to do neck stretch and mouth opening exercises. Telephone follow-up was not provided to usual care group. Furthermore, patients in usual care group went to receive physical therapy were free to do. During the follow-up period, well-trained research nurses (assessors) recorded their physical therapy sections.
- Exercise intervention programs (Experimental): Based on our previous literature review, we will have two major parts of exercises in our intervention: (1) Upper Body Exercise (stretching in shoulder and neck, and mouth-opening); and (2) General Physical Function Training.
  Interventions: Behavioral: Exercise intervention program

INTERVENTIONS:
Behavioral: Exercise intervention program — It was developed, along with usual care, to prevent restricted ROM in both upper body and limited general physical functioning. Patients in exercise intervention group received verbal instructions about stretching major muscles and phsical activity recommendations from a trained nurse (intervenor), and then received the booklet plus DVD.
  The physical therapist who developed and adjusted this program also trained the intervenor. After verifying the intervenor has performed exercise interventions were consistent with the physical therapist, he/she was responsible for all interventions. Therefore, if pain or discomfort persists for more than an hour, the patient should inform the intervenor. The intervention group patients also received telephone follow-up from the intervenor every two weeks until the end of the intervention.
  Arms: Exercise intervention programs

SUMMARY:
Background: Due to the disease location and related treatments in head and neck areas following with concurrent chemoradiation therapy (CCRT), patients might suffer a series of acute distress and limit their physical activities. Limited physical activities might further cause dysfunction in both the upper body and general physical function.

Purposes: This 3-year project will be conducted for three folds, with the purposes to (1) longitudinally examine the upper body function (mouth open abilities/trismus, neck stiffness/flexibility, shoulder function, myofascial pain, and upper arm muscle strengths) and general physical fitness; and (2) develop a 20-week continuous exercise program and test of its effects on improving upper body function, general physical function, fatigue, and quality of life in operable HNC in the first year of being diagnosed as cancer.

Method: The eligible subjects will be newly diagnosed operable HNC patients. For research purpose (1) (Phase 1), we will conduct the data collection for continuous and follow patients for 12 months (Pre-operation, post-op 1, 3, 6, 12 months,/ T1-T5, respectively) for fatigue, upper body function and general physical fitness, and quality of life. A total of 130 subjects are planned to be recruited based on the sample size calculation. For research purpose (2) (Phase 2), from the second year, the 20-week "Multi-Faced Continuous Exercise Program" will be developed and tested in newly diagnosed operable HNC patients, while compare to those standard care control group of their differences in preventing physical dysfunction and increasing physical function for a 20-week period on post-op 1, 3, & 6 months (T0-T2, respectively). Data will be analyzed by both descriptive analysis and the Generalized Estimating Equation (GEE). There will be 130 subjects in each group (N=260 total) based on power analysis principles.

Expected Outcome: The results will increase our knowledge about the changes in physical activities, physical function, and dysfunction; and the levels of the effectiveness of a continuous exercise program on increasing head and neck cancer patients' physical function and quality of life.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNCSCC) is one of the most common cancers in Taiwan. The incidence is rapidly rising and is becoming the leading cause of death in men aged from 40-60 years in recent years. A multimodal treatment approach has led to a relatively good five-year survival rate in HNC patients ranging from 40% to over 50%. A review showed that over the past 10 years, the 5-year survival rate for HNC has increased from 55% to 66%. In other words, with the increasing number of head and neck cancer patients in Taiwan, a rapidly increasing number of survivors and the survival issues related to head and neck cancers are critically necessary to care.

Except those in severe metastasis or terminal condition and those in stage I, the majority of head and neck cancers patients receive a series of treatments, including tumor resection, neck dissection (ND), even reconstruction with free-flap surgery, and CCRT. Due to the disease location and surgery in head and neck areas, many head and neck cancer patients suffer problems in the upper body, particularly head, neck, and shoulder areas. Pain in these areas may cause diminishing function in the upper extremities and weaken the muscle power in the upper extremities.

After the acute distress, patients may also face some long-term problems if those acute problems are not well cared, such as myofascial pain in neck and shoulder areas, trismus from local radiation, and tightness of shoulder. Fatigue and generally declined physical function may also be found to be fatigue, decreasing of physical function, and general malaise. Thus, these declining functions, including both upper extremities and a general weakening in physical function, may further influence patients' physical activities, daily life, and even employment status. It would be therefore very important to systematically assess and intervene in these problems to decrease patients' dysfunction and increase their physical function and quality of life.

Unfortunately, those disease or treatment-related functional declines and decreasing physical activities due to treatments or limited physical conditions may not receive sufficient attention from both health care professionals and patients. Clinically, the major focus has been on treating the life-threatening head and neck cancer, the disease itself. For example, a study was done in UK found that only 8.5% of head and neck cancer survivors reported doing sufficient physical activities which met the current suggested exercise guideline. Very few HNC patients participated in moderate-intensity to vigorous-intensity physical activity. While HNC patients in Taiwan received exercise recommendations before RT, only 16.7% followed WHO exercise recommendations and 14% continued stretching after RT.

Concerning the increasing numbers of head and neck cancer patients and survivors, and the gradually developed physical dysfunction, it would be very important to longitudinally examine the changes of those problems (upper body and general physical function and status of applying physical activities, preferences, and barriers of applying physical activities) during the cancer process. The data would be helpful to develop an evidence-based, brief, easily carried out and comprehensive exercise program that may cover the exercise needs across the cancer process, particularly for the first 6 months of diagnosis (acute treatment phase to off treatment survival phase).

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were adult patients (≥20 years old) with newly diagnosed squamous cell type of HNC patients who received tumor excision and neck dissection (either MRND or SND) within 3-4 weeks
* Part of subjects might with postoperative RT or CCRT

Exclusion Criteria:

* Patients unable to communicate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2013-01-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The 13-item SPADI is composed of two subscales which include pain (5 items), and disability (8 items). The scale is a visual analogue scale, ranging from 0-10 cm, with 0 representing "no difficulty (left anchor)" and 10 representing "so difficult required help (right anchor)". The SPADI total score ranges from 0 to 100 and is obtained by averaging the pain and disability subscale scores. Higher scores indicate greater pain and greater disability. The psychometric testing in a previous study has been reported. The Taiwanese version psychometric testing and scoring in a previous study has been reported.
University of Washington- Quality of Life (UW-QOL) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  University of Washington - Quality of Life (UW-QOL) was characterized of its simplicity and developed to quickly assess head and neck cancer patients' health related QOL. Four versions have been developed since 1993. The current version, UW-QOL version 4 contains 12 items that to assess 12 domains of QOL in head and neck cancer patients. It has been translated into Chinese and tested for its psychometrics in head and neck cancer populations in Taiwan and the 13-item Chinese version (including employment status) of the UWQOL has provided a good reliability and validity.
University of Washington- Quality of Life (UW-QOL) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  University of Washington - Quality of Life (UW-QOL) was characterized of its simplicity and developed to quickly assess head and neck cancer patients' health related QOL. Four versions have been developed since 1993. The current version, UW-QOL version 4 contains 12 items that to assess 12 domains of QOL in head and neck cancer patients. It has been translated into Chinese and tested for its psychometrics in head and neck cancer populations in Taiwan and the 13-item Chinese version (including employment status) of the UWQOL has provided a good reliability and validity.
Hospital Anxiety and Depression Scale (HADS) - Taiwanese version (HADS-Depression subscale) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The 14-item HADS, developed to assess patients' anxiety and depression status, has 7 items that measure anxiety and 7 that measure depression. This scale has been widely used in cancer research to assess patients' psychological distress. The Taiwanese version of HADS has been developed and validated and showed promising psychometrics. In the proposed study, we will use this depression subscale to assess the depression affective dimension of patients' shoulder dysfunction.
Hospital Anxiety and Depression Scale (HADS) - Taiwanese version (HADS-Depression subscale) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The 14-item HADS, developed to assess patients' anxiety and depression status, has 7 items that measure anxiety and 7 that measure depression. This scale has been widely used in cancer research to assess patients' psychological distress. The Taiwanese version of HADS has been developed and validated and showed promising psychometrics. In the proposed study, we will use this depression subscale to assess the depression affective dimension of patients' shoulder dysfunction.
Fatigue Symptom Inventory (FSI) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  We will use the FSI to assess both fatigue intensity (4 items) and fatigue interference (7 items). Psychometric testing of the FSI in cancer patients and healthy subjects showed good validity and reliability. Responses to these items are self-rated on an 11-point Likert-type scale (0=no fatigue at all/no interference; 10=extreme fatigue/extreme interference). The higher the score indicate the greater the levels of fatigue intensity and fatigue interference.
Fatigue Symptom Inventory (FSI) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  We will use the FSI to assess both fatigue intensity (4 items) and fatigue interference (7 items). Psychometric testing of the FSI in cancer patients and healthy subjects showed good validity and reliability. Responses to these items are self-rated on an 11-point Likert-type scale (0=no fatigue at all/no interference; 10=extreme fatigue/extreme interference). The higher the score indicate the greater the levels of fatigue intensity and fatigue interference.
Background Information | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  Data from self-reported demographics (e.g., age and previous exercise behavior) and medical variables (e.g., cancer type, stage, and operation type) were collected.
Background Information | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  Data from self-reported demographics (e.g., age and previous exercise behavior) and medical variables (e.g., cancer type, stage, and operation type) were collected.
Perceived Barriers of Engaging Exercise | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  One open question to report barrier of engaging exercise.
The Karnofsky Performance Status (KPS) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The Karnofsky Performance Status (KPS) scores range from 0 to 100 and has been validated in terms of its reliability and validity.
The Karnofsky Performance Status (KPS) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The Karnofsky Performance Status (KPS) scores range from 0 to 100 and has been validated in terms of its reliability and validity.
Muscle strength | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  Using grip strength meter to measure the strength of right and left upper limbs; and will use microFET 2 to measure the strength of bilateral shoulder-muscle strength (shoulder flexion and horizontal abduction) and hip flexor muscle. Both grip strength meter and microFET 2 provided good reliability and validity for measuring muscle strength in the past studies.
Muscle strength | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  Using grip strength meter to measure the strength of right and left upper limbs; and will use microFET 2 to measure the strength of bilateral shoulder-muscle strength (shoulder flexion and horizontal abduction) and hip flexor muscle. Both grip strength meter and microFET 2 provided good reliability and validity for measuring muscle strength in the past studies.
Cervical range of motion (CROM) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The CROM was measured by using a "CROM device" (Performance Attainment Associates, St Paul, MN, USA). This CROM device has good reliability and validity. The CROM test evaluates the maximum degrees of neck forward flexion, extension, bilateral lateral flexion (right and left), and bilateral rotation (right and left). The procedure begins with warm-up exercises followed by maintaining a neutral position and moving the head naturally and without pain. Measuring two values and calculating the average.
Cervical range of motion (CROM) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The CROM was measured by using a "CROM device" (Performance Attainment Associates, St Paul, MN, USA). This CROM device has good reliability and validity. The CROM test evaluates the maximum degrees of neck forward flexion, extension, bilateral lateral flexion (right and left), and bilateral rotation (right and left). The procedure begins with warm-up exercises followed by maintaining a neutral position and moving the head naturally and without pain. Measuring two values and calculating the average.
Mouth opening | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The normal range of jaw in HNC patients is 3.5. Past research has shown that vernier caliper is reliable tools for measuring mouth openings. The subjects sat upright and measured the distance between the mandibular incisors and the maxilla without feeling pain. Result expressed in centimeters.
Mouth opening | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The normal range of jaw in HNC patients is 3.5. Past research has shown that vernier caliper is reliable tools for measuring mouth openings. The subjects sat upright and measured the distance between the mandibular incisors and the maxilla without feeling pain. Result expressed in centimeters.
  Title:
SF-12 Health Survey (SF-12) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The 12-item SF-12 has eight subscales: physical functioning (2 items), role physical (2 items), role emotional (2 items), mental health (2 items), bodily pain (1 item), general health (1 item), and vitality (1 item), and social functioning (1 item). The SF-12 score include dichotomous items, and three, five-to-six point scales. Each subscale is scored from 0 to 100, with higher scores representing better function.
SF-12 Health Survey (SF-12) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The 12-item SF-12 has eight subscales: physical functioning (2 items), role physical (2 items), role emotional (2 items), mental health (2 items), bodily pain (1 item), general health (1 item), and vitality (1 item), and social functioning (1 item). The SF-12 score include dichotomous items, and three, five-to-six point scales. Each subscale is scored from 0 to 100, with higher scores representing better function.
Brief Pain Inventory - Short Form (BPI-S) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The BPI-S, a self-report scale used to assess patients' pain experience, consists of two major parts, which measure pain intensity and pain interference. The 4-item pain intensity part measures worst pain intensity, pain intensity on average, least pain intensity, and current pain intensity. The 7-item pain interference part assesses the interference of pain on daily life. Each item is rated on a numerical scale from 0 ("no pain at all" or "no interference at all") to 10 ("worst possible pain I can imagine" for pain intensity or "extremely interfering"). The BPI-S has been found to be a reliable and valid measure of pain experience. The Chinese version of BPI-S has also showed promising psychometric characteristics.
Brief Pain Inventory - Short Form (BPI-S) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The BPI-S, a self-report scale used to assess patients' pain experience, consists of two major parts, which measure pain intensity and pain interference. The 4-item pain intensity part measures worst pain intensity, pain intensity on average, least pain intensity, and current pain intensity. The 7-item pain interference part assesses the interference of pain on daily life. Each item is rated on a numerical scale from 0 ("no pain at all" or "no interference at all") to 10 ("worst possible pain I can imagine" for pain intensity or "extremely interfering"). The BPI-S has been found to be a reliable and valid measure of pain experience. The Chinese version of BPI-S has also showed promising psychometric characteristics.
Symptom Severity Scale (SSS) | Phase 1: Change from Baseline (pre-operation) to post-operation 12 months (measured 5 times)
  The SSS is a numeric scale that assesses the severity of common symptoms from 0 (no symptom at all) to 10 (as severe as possible), similar to other numeric rating scales of symptom severity. The SSS has been demonstrated as a reliable scale in cancer-related studies in Taiwan, with satisfactory content validity, face validity, and feasibility. The internal consistency reliability (Cronbach's alpha) ranged from .82 to .91.
Symptom Severity Scale (SSS) | Phase 2: Change from Baseline (post-op 1 month) to post-op 6 months (measured 3 times)
  The SSS is a numeric scale that assesses the severity of common symptoms from 0 (no symptom at all) to 10 (as severe as possible), similar to other numeric rating scales of symptom severity. The SSS has been demonstrated as a reliable scale in cancer-related studies in Taiwan, with satisfactory content validity, face validity, and feasibility. The internal consistency reliability (Cronbach's alpha) ranged from .82 to .91.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — National Taiwan University Hos[ital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601
- [Background] Williams JW Jr, Holleman DR Jr, Simel DL. Measuring shoulder function with the Shoulder Pain and Disability Index. J Rheumatol. 1995 Apr;22(4):727-32. PMID 7791172
- [Background] Yang JL, Lin JJ. Reliability of function-related tests in patients with shoulder pathologies. J Orthop Sports Phys Ther. 2006 Aug;36(8):572-6. doi: 10.2519/jospt.2006.2133. PMID 16915978
- [Background] Hassan SJ, Weymuller EA Jr. Assessment of quality of life in head and neck cancer patients. Head Neck. 1993 Nov-Dec;15(6):485-96. doi: 10.1002/hed.2880150603. PMID 8253555
- [Background] Rogers SN, Scott B, Lowe D. An evaluation of the shoulder domain of the University of Washington quality of life scale. Br J Oral Maxillofac Surg. 2007 Jan;45(1):5-10. doi: 10.1016/j.bjoms.2006.09.007. Epub 2006 Nov 13. PMID 17101200
- [Background] Weymuller EA Jr, Alsarraf R, Yueh B, Deleyiannis FW, Coltrera MD. Analysis of the performance characteristics of the University of Washington Quality of Life instrument and its modification (UW-QOL-R). Arch Otolaryngol Head Neck Surg. 2001 May;127(5):489-93. doi: 10.1001/archotol.127.5.489. PMID 11346422
- [Background] Rogers SN, Gwanne S, Lowe D, Humphris G, Yueh B, Weymuller EA Jr. The addition of mood and anxiety domains to the University of Washington quality of life scale. Head Neck. 2002 Jun;24(6):521-9. doi: 10.1002/hed.10106. PMID 12112548
- [Background] Lee YH, Lai YH, Yueh B, Chu PY, Chen YJ, Chen SC, Wang CP. Validation of the University of Washington Quality of Life Chinese Version (UWQOL-C) for head and neck cancer patients in Taiwan. J Formos Med Assoc. 2017 Apr;116(4):249-256. doi: 10.1016/j.jfma.2017.01.002. Epub 2017 Feb 15. PMID 28214178
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Lampic C, von Essen L, Peterson VW, Larsson G, Sjoden PO. Anxiety and depression in hospitalized patients with cancer: agreement in patient-staff dyads. Cancer Nurs. 1996 Dec;19(6):419-28. doi: 10.1097/00002820-199612000-00002. PMID 8972974
- [Background] Lee Y, Wu YS, Chien CY, Fang FM, Hung CF. Use of the Hospital Anxiety and Depression Scale and the Taiwanese Depression Questionnaire for screening depression in head and neck cancer patients in Taiwan. Neuropsychiatr Dis Treat. 2016 Oct 13;12:2649-2657. doi: 10.2147/NDT.S112069. eCollection 2016. PMID 27789953
- [Background] Chen PY, See LC, Wang CH, Lai YH, Chang HK, & Chen ML. The impact of pain on the anxiety and depression of cancer patients. Formosan Journal of Medicine. 1999; 3: 373-382.
- [Background] Cheng PT, Hao SP, Lin YH, Yeh AR. Objective comparison of shoulder dysfunction after three neck dissection techniques. Ann Otol Rhinol Laryngol. 2000 Aug;109(8 Pt 1):761-6. doi: 10.1177/000348940010900811. PMID 10961810
- [Background] Hsu C, Shen YC, Cheng CC, Hong RL, Chang CJ, Cheng AL. Difference in the incidence trend of nasopharyngeal and oropharyngeal carcinomas in Taiwan: implication from age-period-cohort analysis. Cancer Epidemiol Biomarkers Prev. 2006 May;15(5):856-61. doi: 10.1158/1055-9965.EPI-05-0821. PMID 16702360
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Shun SC, Beck SL, Pett MA, Berry PH. Psychometric testing of three Chinese fatigue instruments in Taiwan. J Pain Symptom Manage. 2006 Aug;32(2):155-67. doi: 10.1016/j.jpainsymman.2006.02.011. PMID 16877183
- [Background] Karnofsky D. Performance scale. Factors that influence the therapeutic response in cancer: a comprehensive treatise. Plenum Press, New York; 1977.
- [Background] Schag CC, Heinrich RL, Ganz PA. Karnofsky performance status revisited: reliability, validity, and guidelines. J Clin Oncol. 1984 Mar;2(3):187-93. doi: 10.1200/JCO.1984.2.3.187. PMID 6699671
- [Background] Schaubert KL, Bohannon RW. Reliability and validity of three strength measures obtained from community-dwelling elderly persons. J Strength Cond Res. 2005 Aug;19(3):717-20. doi: 10.1519/R-15954.1. PMID 16095431
- [Background] Williams MA, McCarthy CJ, Chorti A, Cooke MW, Gates S. A systematic review of reliability and validity studies of methods for measuring active and passive cervical range of motion. J Manipulative Physiol Ther. 2010 Feb;33(2):138-55. doi: 10.1016/j.jmpt.2009.12.009. PMID 20170780
- [Background] Norkin CC, White DJ. Measurement Of Joint Motion: A Guide To Goniometry: F.A. Davis Company; 2016.
- [Background] Dijkstra PU, Huisman PM, Roodenburg JL. Criteria for trismus in head and neck oncology. Int J Oral Maxillofac Surg. 2006 Apr;35(4):337-42. doi: 10.1016/j.ijom.2005.08.001. Epub 2005 Nov 8. PMID 16280237
- [Background] Best N, Best S, Loudovici-Krug D, Smolenski UC. Measurement of mandible movements using a vernier caliper--an evaluation of the intrasession-, intersession- and interobserver reliability. Cranio. 2013 Jul;31(3):176-80. doi: 10.1179/crn.2013.028. PMID 23971158
- [Background] Johnson DE, Burtness B, Leemans CR, Lui VWY, Bauman JE, Grandis JR. Head and neck squamous cell carcinoma. Nat Rev Dis Primers. 2020 Nov 26;6(1):92. doi: 10.1038/s41572-020-00224-3. PMID 33243986
- [Background] World Health Organization [WHO]. Locally advanced squamous carcinoma of the head and neck. 2014. Retrieved from https://www.who.int/selection_medicines/committees/expert/20/applications/HeadNeck.pdf
- [Background] Health Promotion Administration Ministry of Health And Welfare [HPA] ROC. 2017 Cancer registry annual report in Taiwan. 2019. Retrieved from https://www.hpa.gov.tw/Pages/Detail.aspx?nodeid=269&pid=12235
- [Background] Crozier E, Sumer BD. Head and neck cancer. Med Clin North Am. 2010 Sep;94(5):1031-46. doi: 10.1016/j.mcna.2010.05.014. PMID 20736111
- [Background] Carr SD, Bowyer D, Cox G. Upper limb dysfunction following selective neck dissection: a retrospective questionnaire study. Head Neck. 2009 Jun;31(6):789-92. doi: 10.1002/hed.21018. PMID 19260131
- [Background] Umeda M, Shigeta T, Takahashi H, Oguni A, Kataoka T, Minamikawa T, Shibuya Y, Komori T. Shoulder mobility after spinal accessory nerve-sparing modified radical neck dissection in oral cancer patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jun;109(6):820-4. doi: 10.1016/j.tripleo.2009.11.027. Epub 2010 Mar 17. PMID 20299249
- [Background] van Wilgen CP, Dijkstra PU, van der Laan BF, Plukker JT, Roodenburg JL. Shoulder and neck morbidity in quality of life after surgery for head and neck cancer. Head Neck. 2004 Oct;26(10):839-44. doi: 10.1002/hed.20052. PMID 15390203
- [Background] Stuiver MM, van Wilgen CP, de Boer EM, de Goede CJ, Koolstra M, van Opzeeland A, Venema P, Sterken MW, Vincent A, Dijkstra PU. Impact of shoulder complaints after neck dissection on shoulder disability and quality of life. Otolaryngol Head Neck Surg. 2008 Jul;139(1):32-9. doi: 10.1016/j.otohns.2008.03.019. PMID 18585558
- [Background] van Wilgen CP, Bloten H, Oeseburg B. Results of a multidisciplinary program for patients with fibromyalgia implemented in the primary care. Disabil Rehabil. 2007 Aug 15;29(15):1207-13. doi: 10.1080/09638280600949860. PMID 17653994
- [Background] Eades M, Chasen M, Bhargava R. Rehabilitation: long-term physical and functional changes following treatment. Semin Oncol Nurs. 2009 Aug;25(3):222-30. doi: 10.1016/j.soncn.2009.05.006. PMID 19635401
- [Background] Luctkar-Flude M, Groll D, Woodend K, Tranmer J. Fatigue and physical activity in older patients with cancer: a six-month follow-up study. Oncol Nurs Forum. 2009 Mar;36(2):194-202. doi: 10.1188/09.ONF.194-202. PMID 19273408
- [Background] Rogers LQ, Courneya KS, Robbins KT, Malone J, Seiz A, Koch L, Rao K, Nagarkar M. Physical activity and quality of life in head and neck cancer survivors. Support Care Cancer. 2006 Oct;14(10):1012-9. doi: 10.1007/s00520-006-0044-7. Epub 2006 Mar 15. PMID 16538497
- [Background] Rogers SN, Lowe D, Yueh B, Weymuller EA Jr. The physical function and social-emotional function subscales of the University of Washington Quality of Life Questionnaire. Arch Otolaryngol Head Neck Surg. 2010 Apr;136(4):352-7. doi: 10.1001/archoto.2010.32. PMID 20403851
- [Background] Campana JP, Meyers AD. The surgical management of oral cancer. Otolaryngol Clin North Am. 2006 Apr;39(2):331-48. doi: 10.1016/j.otc.2005.11.005. PMID 16580915
- [Background] Fang YY, Wang CP, Chen YJ, Lou PJ, Ko JY, Lin JJ, Chen MR, Lai YH. Physical activity and fitness in survivors of head and neck cancer. Support Care Cancer. 2021 Nov;29(11):6807-6817. doi: 10.1007/s00520-021-06192-y. Epub 2021 May 17. PMID 33997941
- [Background] Liao CT, Wang HM, Chang JT, Ng SH, Hsueh C, Lee LY, Lin CH, Chen IH, Huang SF, Yen TC. Analysis of risk factors for distant metastases in squamous cell carcinoma of the oral cavity. Cancer. 2007 Oct 1;110(7):1501-8. doi: 10.1002/cncr.22959. PMID 17868119
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Cleeland CS. Measurement and prevalence of pain in cancer. Semin Oncol Nurs. 1985 May;1(2):87-92. doi: 10.1016/s0749-2081(85)80041-3. No abstract available. PMID 3849841
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Lai YH, Guo SL, Keefe FJ, Tsai SL, Chien CC, Sung YC, Chen ML. Effects of brief pain education on hospitalized cancer patients with moderate to severe pain. Support Care Cancer. 2004 Sep;12(9):645-52. doi: 10.1007/s00520-004-0626-1. PMID 15127282
- [Background] Lai YH. Symptom distress and home care needs in patients receiving chemotherapy in an outpatient setting. Journal of Nursing Research (Chinese). 1998; 6:279-289.
- [Background] Chen SC, Lai YH, Liao CT, Lin CC, Chang JT. Changes of symptoms and depression in oral cavity cancer patients receiving radiation therapy. Oral Oncol. 2010 Jul;46(7):509-13. doi: 10.1016/j.oraloncology.2010.02.024. Epub 2010 Mar 21. PMID 20308004
- [Background] Chen SC, Lai YH, Liao CT, Chang JT, Lin CY, Fan KH, Huang BS. Supportive care needs in newly diagnosed oral cavity cancer patients receiving radiation therapy. Psychooncology. 2013 Jun;22(6):1220-8. doi: 10.1002/pon.3126. Epub 2012 Jun 25. PMID 22730021